CLINICAL TRIAL: NCT01127802
Title: Changes of Functional Status, Symptoms Distress and Quality of Life in Patients Undergoing CABG Surgery
Brief Title: Changes of Functional Status, Symptoms Distress and Quality of Life in Patients Undergoing Coronary Artery Bypass Graft (CABG) Surgery
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Cheryl Chia-Hui Chen, Department of Nursing, College of Medicine, National Taiwan University
Other Study IDs: 201003017R
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2010-05-21 (Estimated); Status verified 2010-05

CONDITIONS: Coronary Artery Bypass Graft Surgery
Keywords: CABG; functional status; symptoms distress; quality of life; the trajectory of functional status; the changes of symptoms distress; the changes of quality of life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to explore the changes of functional status, symptoms distress and quality of life in patients undergoing coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
This is an observational cohort study. The participants will be inpatients undergoing elective CABG surgery at one tertiary medical center. Functional status (including activity of daily living, cognitive and nutritional status), symptom distress, and quality of life will be measured at multiple points: pre-surgery, day 1 to 7 post-surgery, before discharge, and 2-4 weeks after discharge. Structured questionnaire will be used to collect demographic and medical characteristics. The Barthel Index, hand-held dynamometer, 6-minute walking test, Mini-Nutritional Assessment (MNA), Mini-Mental State Examination (MMSE), Confusion Assessment Method (CAM), Symptoms Distress Scale, and Short-Form-36 Health Survey (SF-36) will be used to collect functional data and compared for changes. The trajectory of functional status, symptoms distress, and quality of life will be further analyzed. The findings will add to the literature by raising the awareness on changes of functional status, symptoms distress, and quality of life for patients undergoing elective CABG so targeted and timely intervention could be developed and planned.

ELIGIBILITY:
Inclusion Criteria:

* receive elective coronary artery bypass surgery
* able to communicate in Chinese and Taiwanese
* walk independently or use walker
* length of stay is over 7 days

Exclusion Criteria:

* unable to walk
* mechanical ventilation
* neural or muscle disease to influence ambulation(ex: Parkinson Disease)
* asthma
* severe psychotic disorder that prevents patient from participating in test

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients undergoing elective CABG surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-03 (Estimated); Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Hui Chen, Ph. D., Study Chair — National Taiwan University Hospital